CLINICAL TRIAL: NCT03079687
Title: A Multiple Patient Expanded Access Program for Olaparib Tablets for the Maintenance Treatment Following Response (Complete Response or Partial Response) to Platinum-based Chemotherapy in Patients With Platinum-sensitive Relapsed High-grade Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer.
Brief Title: Expanded Access Program for Olaparib Tablets as Maintenance Therapy in Patients With Ovarian, Fallopian Tube or Primary Peritoneal Cancer.
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816R00014
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; gynaecological cancer; platinum-sensitive disease; platinum-sensitive relapsed; Olaparib; Ovarian Neoplasms; Neoplasms; Ovarian Disease; fallopean tube cancer; primary peritoneal cancer; epithelial ovarian cancer; PARP inhibitors; Poly (ADP-ribose) polymerase inhibitors.
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Ovarian Diseases; Carcinoma, Ovarian Epithelial | interventions — olaparib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Olaparib tablets — Patients will receive olaparib tablets 300mg (two 150mg tablets) twice daily.

SUMMARY:
This is an open-label, single-arm, international, multicenter Multiple Patient Expanded Access Program (MPEAP). The program is designed to provide treatment access to olaparib tablets for patients with platinum-sensitive relapsed high-grade epithelial ovarian, fallopian tube or primary peritoneal cancer without other treatment options or eligible for an olaparib clinical trials.

DETAILED DESCRIPTION:
The Multiple Patient Expanded Access Program is designed to provide treatment access to olaparib tablets for patients with platinum-sensitive relapsed high-grade epithelial ovarian, fallopian tube or primary peritoneal cancer who are in response (complete response or partial response) following platinum-based chemotherapy. The dose of olaparib tablets is 300 mg (two 150 mg tablets) taken twice daily, equivalent to a total daily dose of 600 mg. The 100 mg tablet is available for dose reduction. Treatment may continue until disease progression, unacceptable toxicity or withdrawal of patient consent. The program will collect observational data only.

ELIGIBILITY:
Inclusion criteria

For inclusion in the program patients must fulfill the following criteria:

* Provision of informed consent prior to any program specific procedures
* Female patients ≥ 18 years of age and has platinum-sensitive relapsed high grade epithelial ovarian, primary peritoneal or fallopian tube cancer
* Patient is in response (complete response or partial response) following platinum-based chemotherapy.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of program treatment.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential.

Exclusion criteria:

Patients should not enter the program if any of the following exclusion criteria are fulfilled:

* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors.
* Concomitant use of known strong or moderate CYP3A inducers. The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patient with moderate or severe hepatic impairment.
* Breast feeding women.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Research Site, Duarte, California
  - Research Site, Newport Beach, California
  - Research Site, Roseville, California
  - Research Site, Gainesville, Florida
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon